CLINICAL TRIAL: NCT02943018
Title: Interobserver Agreement in Perineal Ultrasound of the Anovaginal Distance- a Methodology-study
Brief Title: Anovaginal Distance, Interobserver Agreement
Status: Completed | Type: Observational
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Eva Uustal, Senior consultant, Ostergotland County Council, Sweden
Other Study IDs: OstergotlandCCAVD
Record Dates: First submitted 2016-10-18; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Pelvic Floor Disorders
Keywords: ultrasound anovaginal distance, observer variation
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- anovaginal distance variation: 3 measurements
  Interventions: Other: anovaginal distance variation

INTERVENTIONS:
Other: anovaginal distance variation — Kappa calculation

SUMMARY:
Interobserver variation in measuring the anovaginal distance (AVD) with perineal ultrasound

DETAILED DESCRIPTION:
Aims: This study describes perineal ultrasound measurement of the AVD in regard to ease of learning and interobserver agreement, in order to establish if the method is reliable to use in further research about objective postpartum description of perineal tears.

Methods: To educate the examiners, the method was shown and described by an experienced examiner. The examiners then measured the anovaginal distance in one woman repeatedly with until similar results (+/- 5 mm ) were achieved. The woman was in the lithotomy position and a vaginal ultrasound probe was used. The AVD in another 40 women was then measured and documented by two examiners, right after the other, who were blinded to the other´s results. The distance was measured between the mucosal margin of the internal anal sphincter and the vaginal probe. Interobserver agreement was calculated using Kappa-score.

ELIGIBILITY:
Inclusion Criteria:

Examiners; the gynecologists authoring the study

Patients:

* any women visiting the gynaecological outpatient clinic of Linköping University Hospital where a vaginal ultrasound examination was performed

Exclusion Criteria:

Examiners: n/a

Patients:

* inability to understand spoken or written Swedish

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The examiners whose measurements were compared for interobserver varialility were gynecologists working inte the department.
  The study population to perform measurements on was recruited from women visiting the gynaecological outpatient clinic of Linköping University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
interobserver variation in measurements of the anovaginal distance with perineal ultrasound | immediate
  3 measurements per investigator and patient, comparing variation, using kappa value

SECONDARY OUTCOMES:
Ease of learning the technique of perineal ultrasound to measure the anovaginal distance | immediate
  how many measurements did the investigator learning the procedure need to perform produce a measurement that was within 5 mm of the measurements of the teacher

CONTACTS AND LOCATIONS:
Overall Officials: Marie I Blomberg, MD PhD, Principal Investigator — head of department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faltin DL, Boulvain M, Floris LA, Irion O. Diagnosis of anal sphincter tears to prevent fecal incontinence: a randomized controlled trial. Obstet Gynecol. 2005 Jul;106(1):6-13. doi: 10.1097/01.AOG.0000165273.68486.95. PMID 15994610
- [Background] Starck M, Bohe M, Fortling B, Valentin L. Endosonography of the anal sphincter in women of different ages and parity. Ultrasound Obstet Gynecol. 2005 Feb;25(2):169-76. doi: 10.1002/uog.1818. PMID 15685668
- [Background] Andrews V, Sultan AH, Thakar R, Jones PW. Occult anal sphincter injuries--myth or reality? BJOG. 2006 Feb;113(2):195-200. doi: 10.1111/j.1471-0528.2006.00799.x. PMID 16411998
- [Background] Peschers UM, DeLancey JO, Schaer GN, Schuessler B. Exoanal ultrasound of the anal sphincter: normal anatomy and sphincter defects. Br J Obstet Gynaecol. 1997 Sep;104(9):999-1003. doi: 10.1111/j.1471-0528.1997.tb12056.x. PMID 9307524
- [Background] Poen AC, Felt-Bersma RJ, Cuesta MA, Meuwissen GM. Vaginal endosonography of the anal sphincter complex is important in the assessment of faecal incontinence and perianal sepsis. Br J Surg. 1998 Mar;85(3):359-63. doi: 10.1046/j.1365-2168.1998.00616.x. PMID 9529493
- [Background] Stewart LK, Wilson SR. Transvaginal sonography of the anal sphincter: reliable, or not? AJR Am J Roentgenol. 1999 Jul;173(1):179-85. doi: 10.2214/ajr.173.1.10397123.
- [Background] Frudinger A, Bartram CI, Kamm MA. Transvaginal versus anal endosonography for detecting damage to the anal sphincter. AJR Am J Roentgenol. 1997 Jun;168(6):1435-8. doi: 10.2214/ajr.168.6.9168703.
- [Background] Timor-Tritsch IE, Monteagudo A, Smilen SW, Porges RF, Avizova E. Simple ultrasound evaluation of the anal sphincter in female patients using a transvaginal transducer. Ultrasound Obstet Gynecol. 2005 Feb;25(2):177-83. doi: 10.1002/uog.1827. PMID 15660445
- [Background] Yang SH, Huang WC, Yang SY, Yang E, Yang JM. Validation of new ultrasound parameters for quantifying pelvic floor muscle contraction. Ultrasound Obstet Gynecol. 2009 Apr;33(4):465-71. doi: 10.1002/uog.6338. PMID 19306473
- [Background] Olsen IP, Wilsgaard T, Kiserud T. Transvaginal three-dimensional ultrasound: a method of studying anal anatomy and function. Ultrasound Obstet Gynecol. 2011 Mar;37(3):353-60. doi: 10.1002/uog.8873. PMID 21337656
- [Background] Valsky DV, Messing B, Petkova R, Savchev S, Rosenak D, Hochner-Celnikier D, Yagel S. Postpartum evaluation of the anal sphincter by transperineal three-dimensional ultrasound in primiparous women after vaginal delivery and following surgical repair of third-degree tears by the overlapping technique. Ultrasound Obstet Gynecol. 2007 Feb;29(2):195-204. doi: 10.1002/uog.3923. PMID 17219371
- [Background] Shobeiri SA, White D, Quiroz LH, Nihira MA. Anterior and posterior compartment 3D endovaginal ultrasound anatomy based on direct histologic comparison. Int Urogynecol J. 2012 Aug;23(8):1047-53. doi: 10.1007/s00192-012-1721-3. Epub 2012 Mar 9. PMID 22402641
- [Background] Falkert A, Willmann A, Endress E, Meint P, Seelbach-Gobel B. Three-dimensional ultrasound of pelvic floor: is there a correlation with delivery mode and persisting pelvic floor disorders 18-24 months after first delivery? Ultrasound Obstet Gynecol. 2013 Feb;41(2):204-9. doi: 10.1002/uog.11214. PMID 22745047
- [Background] Santoro GA, Shobeiri SA, Petros PP, Zapater P, Wieczorek AP. Perineal body anatomy seen by three-dimensional endovaginal ultrasound of asymptomatic nulliparae. Colorectal Dis. 2016 Apr;18(4):400-9. doi: 10.1111/codi.13119. PMID 26382090
- [Background] Sultan AH, Loder PB, Bartram CI, Kamm MA, Hudson CN. Vaginal endosonography. New approach to image the undisturbed anal sphincter. Dis Colon Rectum. 1994 Dec;37(12):1296-9. doi: 10.1007/BF02257800. PMID 7995162
- [Background] Larson KA, Yousuf A, Lewicky-Gaupp C, Fenner DE, DeLancey JO. Perineal body anatomy in living women: 3-dimensional analysis using thin-slice magnetic resonance imaging. Am J Obstet Gynecol. 2010 Nov;203(5):494.e15-21. doi: 10.1016/j.ajog.2010.06.008. PMID 21055513
- [Background] Uustal Fornell, E. The perineal body thickness - normal values and correlation to pelvic floor dysfunction. Abstract 344, IUGA 2005
- [Background] Hall RJ, Rogers RG, Saiz L, Qualls C. Translabial ultrasound assessment of the anal sphincter complex: normal measurements of the internal and external anal sphincters at the proximal, mid-, and distal levels. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Aug;18(8):881-8. doi: 10.1007/s00192-006-0254-z. Epub 2007 Jan 13. PMID 17221149
- [Background] Viera AJ, Garrett JM. Understanding interobserver agreement: the kappa statistic. Fam Med. 2005 May;37(5):360-3. PMID 15883903
- [Background] Santoro GA, Wieczorek AP, Shobeiri SA, Mueller ER, Pilat J, Stankiewicz A, Battistella G. Interobserver and interdisciplinary reproducibility of 3D endovaginal ultrasound assessment of pelvic floor anatomy. Int Urogynecol J. 2011 Jan;22(1):53-9. doi: 10.1007/s00192-010-1233-y. Epub 2010 Aug 11. PMID 20700728
- [Background] Zetterstrom JP, Mellgren A, Madoff RD, Kim DG, Wong WD. Perineal body measurement improves evaluation of anterior sphincter lesions during endoanal ultrasonography. Dis Colon Rectum. 1998 Jun;41(6):705-13. doi: 10.1007/BF02236256. PMID 9645738
- [Background] Ozyurt S, Aksoy H, Gedikbasi A, Yildirim G, Aksoy U, Acmaz G, Ark C. Screening occult anal sphincter injuries in primigravid women after vaginal delivery with transperineal use of vaginal probe: a prospective, randomized controlled trial. Arch Gynecol Obstet. 2015 Oct;292(4):853-9. doi: 10.1007/s00404-015-3708-z. Epub 2015 Apr 10. PMID 25859828
- [Result] Faltin DL, Boulvain M, Stan C, Epiney M, Weil A, Irion O. Intraobserver and interobserver agreement in the diagnosis of anal sphincter tears by postpartum endosonography. Ultrasound Obstet Gynecol. 2003 Apr;21(4):375-7. doi: 10.1002/uog.86. PMID 12704747